CLINICAL TRIAL: NCT04139785
Title: Moodbuster, a Guided Self-help Intervention for Prevention of Depression in Primary Care
Brief Title: An Online Self-help Intervention for Prevention of Depression in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mental Health Foundation, London (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); VU University of Amsterdam (Other); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0001
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Depression
Keywords: Depression; Anxiety; Prevention; Public Mental Health; Primary Care
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study will follow a two-armed randomised controlled, single-blind, parallel group, wait-list control design. Individuals with mild-moderate symptoms of depression who do not have a diagnosis of depression are invited to participate
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Guided Cognitive Behavioural Therapy based app
  Interventions: Other: Moodbuster
- Care as usual (No Intervention): Care as usual

INTERVENTIONS:
Other: Moodbuster — Moodbuster intervention comprises three elements: (1) a web-based interface providing the patients access to CBT therapies, (2) a web-based portal for the trial co-ordinator and researchers, where they can view participation, amend modules and send login codes, (3) a mobile phone component which enables daily EMA monitoring of mood state, cognitions, activities, social interaction, and sleep.
  The mobile application will be used to capture EMA data.
  Arms: Intervention

SUMMARY:
Depression is a common condition and is the leading cause of disability worldwide. Preventing or delaying the onset of depression is an important way to reduce the burden of depression. Some research suggests online methods may be effective in preventing depression, but to date, few studies have looked at the application of these methods in the UK.

This study aims to assess the effects of an online self-help intervention (Moodbuster) on preventing depression in a primary care population, who are experiencing mild-moderate symptoms of depression, but do not meet the threshold for diagnosis.

A randomised control design with a six-month and nine-month follow up will be used to compare Moodbuster to a wait-listed control group. Then, a qualitative process evaluation will be used to understand the barriers and facilitators of implementing the intervention.

Eligible participants in Greater Manchester (individuals with mild to moderate symptoms of depression, who do not have a diagnosis of major depressive disorder and have access to the internet) will take part in a 6-week online self-help programme, accompanied by three telephone calls with a trained researcher to support them in their use of the programme. Researchers will follow-up with participants six and nine months after starting the programme to measure depression, anxiety, quality of life, and use of services. The process evaluation will involve qualitative interviews with participants and focus groups with practitioners who referred individuals to the study.

This study will assess the effects of Moodbuster on preventing depression and barriers and facilitators of implementing such an intervention in a UK primary care population. It is hypothesised that the intervention group will display reduced depression symptoms and incidence, reduced service use, and improved quality of life, and the intervention will be acceptable to a UK primary care population.

DETAILED DESCRIPTION:
Depression is a common, often recurring, condition and the leading cause of disability worldwide. In the UK, the one-week prevalence of depression is estimated at 3.3%, and by 2026, the cost of depression to the UK economy is estimated to reach £12.15 billion in lost earnings and service use costs. There are two main strategies to reduce the burden of depression, treatment and prevention. Treatment for depression is, even with full coverage of services to all those who need it, not enough.to avert the total burden of disease. Indeed, whist treatment is crucial, even if all people with depression received evidence-based treatment, it is likely that only 35% of the burden (years lived with disabilities) would be averted. Prevention strategies are an integral part of reducing the burden of depression through fully preventing, or otherwise delaying, its onset. One way to improve the reach of prevention interventions and to deliver such approaches at scale is to offer interventions via digital technologies such as websites, computer programmes, or apps. This allows for a larger reach and it may help reach communities which are currently under-served by traditional mental health services. Whilst digital tools have been shown to be effective and acceptable in primary care for the treatment of depression, less research has been conducted on its effectiveness or barriers and facilitators to implementation for prevention. A 2017 meta-analysis identified ten trials on the effectiveness of digital interventions for the prevention of anxiety and depression. The review found promising evidence for the use of digital interventions for prevention, finding a small but positive effect on depression symptoms in the short-term (0.25, [0.09-0.41], p = 0.003). However, the majority of these studies were conducted outside of the UK, in Germany, Australia, USA, Japan, Norway, and the Netherlands. The trials also represented a mix of universal interventions, and indicated/selective efforts targeted to university students, older adults, and young adults. Of the two studies identified that were conducted in the UK, both had a short-term follow up, one of 6 weeks, and the other 12 weeks and did not include diagnostic outcome assessments. This suggests there is still more to learn about the application of digital technologies in the UK for the prevention of depression, and the medium to longer term effects of such interventions.

Research questions:

1. Can an online self-help tool reduce depression symptoms and help support the prevention of depression?
2. What are the effects of Moodbuster on the development of depression, anxiety symptoms, quality of life, and service use, and are there any negative unintended effects?
3. What are the barriers and facilitators to implementing an online tool for prevention in primary care and community settings?

Research hypothesis:

It is hypothesised that the intervention group will display reduced depression symptoms and incidence, reduced service use, and improved quality of life, and the intervention will be acceptable to a UK primary care population.

Recruitment:

Participants will be recruited via three routes:

1. Direct referral from GPs in participating practices, who feel the study would be appropriate for their patients
2. Through a software tool (FARSITE) that allows for the secure searching of GP records for potential study participants at participating GP practices
3. Self-referral by individuals in response to recruitment campaign launched both in-print and online by the Mental Health Foundation (MHF).

The final sample of participants accepted for the trial will be randomly allocated to either the intervention arm or the Treatment as Usual (TAU) arm by an independent statistician based at the University of Manchester.

Intervention:

Those assigned to the intervention will take part in a six-week online self-help programme called Moodbuster. Use of the programme will be supported by three telephone calls from a trained researcher at baseline, three weeks, and six weeks. The calls will serve to support participants with their use of Moodbuster and resolve any technical issues. Treatment as usual during the study period will involve participants carrying on as they ordinarily would and seeking support as and when they feel it is needed using the (clinical) resources and services available in their area. Those assigned to the TAU arm will receive the stand-alone online intervention for free after the nine-month study period and will have access for an additional 9 months.

Data Collection:

Baseline data will be collected via online questionnaires, and an interview. Participants in the intervention arm will be asked to complete a second set of online questionnaires upon completing the six-week self-help programme. This will involve the same set of online questionnaires completed at baseline with additional items related to acceptability of the self-help programme. Participants in both groups will be contacted again at six months and nine months for follow-up data collection, which will involve the same set of online questionnaires that were completed at baseline. At nine months, participants will also be asked to participate in a second diagnostic telephone interview with trained researchers. Sub-groups of participants taking part in the intervention arm of the study will be selected for inclusion in the qualitative process evaluation. The aim is to recruit 20-25 participants for interview. In depth semi-structured interviews will be conducted with participants one month after the end of the intervention. Participants will be asked questions related to barriers and facilitators encountered in the use of Moodbuster, the perceived impact of Moodbuster on their daily lives, and their motivations for taking part in the study. Interviews will last approximately 30 minutes and will be conducted by study team researchers over the phone. Additional focus groups will be conducted with primary care professionals involved in the recruitment and referral to the intervention. Purposive sampling will be used to select staff to reflect different areas of expertise. Focus groups will be conducted one month after the end of the intervention and will explore professionals' perspectives on the implementation of the intervention. This will include the perceived impact of the tool and barriers and facilitators to use.

Sample size: Intervention

For our design, which assesses baseline and two follow-up measurements, we anticipate an effect size of 0.30 at nine-month. This estimate is based on prior meta-analyses on depression prevention.

An effect size of 0.30 indicates a sample size of N = 116 per arm, or N = 232 for the full trial. Accounting for 20% drop-out, we would require a sample size of N = 290 participants. This is based on the assumption that the correlation between baseline and follow-up is 0.5.

Sub-Sample Size: Process evaluation

For the qualitative component, we will aim to recruit up to 25 participants for interviews, and a further 15 professionals for focus groups. This number ensures sufficient data to answer the research questions and is achievable within the timescales of the project. It is consistent with previous research applying thematic analysis to interview data in mental health. The exact number of participants recruited will depend on the richness of the interview data and whether new themes continue to emerge. Recruitment and data collection will continue until collection of new data does not shed any further light on the issue under investigation and saturation has been reached.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above
* Willing and able to give informed consent for participation
* Have sub-threshold mild to moderate symptoms of depression (PHQ-9 scores of 5-9)
* Access to the internet
* In possession of a mobile smartphone (Android) and computer
* In possession of an e-mail address

Exclusion Criteria:

* Currently, or has ever, met DSM-IV criteria for major depression, bipolar disorder, substance dependence, or a psychotic disorder
* Has had a major depressive episode (meeting DSM-IV criteria) as measured by the BDI-II
* Is currently receiving psychotherapy, on a waiting list for psychotherapy, or received psychotherapy in the last six months for any mental health problem
* Is unable to speak, read, or write in English
* Has started a course of antidepressants within the last six weeks
* Endorsement of PHQ item 9 "thoughts you would be better off dead, or of hurting yourself in some way"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Depression Symptoms (Patient Health Questionnaire, 9-item) | 6 months
  Difference in self-reported depression symptoms between intervention and control groups. The PHQ-9 is formed of nine items, each item is scored from 0-3 (0 = not at all; 3 = nearly every day) yielding a total score between 0 and 27. Higher scores are associated with decreased functional status and increased symptom-related difficulties.
Depression Symptoms (Patient Health Questionnaire, 9-item) | 9 months
  Difference in self-reported depression symptoms between intervention and control groups. The PHQ-9 is formed of nine items, each item is scored from 0-3 (0 = not at all; 3 = nearly every day) yielding a total score between 0 and 27. Higher scores are associated with decreased functional status and increased symptom-related difficulties.

SECONDARY OUTCOMES:
Depression Onset (Beck Depression Inventory-II) | 9 months
  Onset of depression considered as a survival outcome for control compared to intervention group.Higher scores indicate greater symptom severity. In non-clinical populations, scores above 20 indicate depression.
Anxiety Symptoms (Generalised Anxiety Disorder Assessment, 7-item) | 6 months
  Difference in self-reported anxiety symptoms between intervention and control groups. The GAD-7 is composed of seven items, each item is scored from 0-3 (0 = not at all; 3 = nearly every day), yielding a total score between 0 and 21. Scores of 5, 10 and 15 are considered as the cut-off points for mild, moderate and severe anxiety.
Anxiety Symptoms (Generalised Anxiety Disorder Assessment, 7-item) | 9 months
  Difference in self-reported anxiety symptoms between intervention and control groups. The GAD-7 is composed of seven items, each item is scored from 0-3 (0 = not at all; 3 = nearly every day), yielding a total score between 0 and 21. Scores of 5, 10 and 15 are considered as the cut-off points for mild, moderate and severe anxiety.
Quality of Life (EQ-5D-5L) | 6 months
  Difference in self-reported quality of life between intervention and control group as measured by the EQ-5D-5L. This is a five item questionnaire which asks about Mobility, Self-Care, Usual Activities, Pain Discomfort and Anxiety/Depression. The index score ranges from less than zero which indicates the patient rates their health related quality of life as "worse than dead", to one which indicates full heath.
Quality of Life (EQ-5D-5L) | 9 months
  Difference in self-reported quality of life between intervention and control group as measured by the EQ-5D-5L. This is a five item questionnaire which asks about Mobility, Self-Care, Usual Activities, Pain Discomfort and Anxiety/Depression. The index score ranges from less than zero which indicates the patient rates their health related quality of life as "worse than dead", to one which indicates full heath.
Intervention Acceptability (Client Satisfaction Questionnaire, 8-item) | Post-Intervention (6 weeks from date of randomization)
  Overall self-reported satisfaction with intervention (for intervention group) as measured by the CSQ-8. Scores range from 8 to 32 with higher scores indicating higher satisfaction.
Negative Effects of Intervention (Inventory for Negative Effects of Psychotherapy) | Post-Intervention (6 weeks from date of randomization)
  Overall self-reported negative effects of intervention as measured by the INEP (for intervention group only). This measure consists of 15 items dealing with the potential side effects of psychotherapy. Items are scared on a 4-point Likert scale with low scores indicating negative effects of therapy and high scores indicating positive effects of psychotherapy.
Barriers and Facilitators to Intervention Use (Qualitative) | Post-Intervention (10 weeks from date of randomization)
  Themes emerging from qualitative interviews with intervention group participants.
Changes in mood, rumination, sleep, and esteem (Ecological Momentary Assessments) | Once per day for duration of intervention (period of 6 weeks from date of randomization)
  Changes in ratings of mood (for intervention group only) for duration of intervention rated on a visual analogue scale. Higher ratings indicate better mood, rumination, quality of sleep and higher levels of esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M Abel, PhD, Principal Investigator — University of Manchester; Antonis Kousoulis, MD, Study Director — Mental Health Foundation
Locations (1):
- University of Manchester, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
To share with other researchers, upon request, anonymised and encrypted individual patient data that underlies results from any resulting academic publications.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Six months through 10 years following publication.

REFERENCES:
- [Background] Buntrock C, Ebert DD, Lehr D, Smit F, Riper H, Berking M, Cuijpers P. Effect of a Web-Based Guided Self-help Intervention for Prevention of Major Depression in Adults With Subthreshold Depression: A Randomized Clinical Trial. JAMA. 2016 May 3;315(17):1854-63. doi: 10.1001/jama.2016.4326. PMID 27139058
- [Background] Chisholm D, Sweeny K, Sheehan P, Rasmussen B, Smit F, Cuijpers P, Saxena S. Scaling-up treatment of depression and anxiety: a global return on investment analysis. Lancet Psychiatry. 2016 May;3(5):415-24. doi: 10.1016/S2215-0366(16)30024-4. Epub 2016 Apr 12. PMID 27083119
- [Background] Ustun TB, Ayuso-Mateos JL, Chatterji S, Mathers C, Murray CJ. Global burden of depressive disorders in the year 2000. Br J Psychiatry. 2004 May;184:386-92. doi: 10.1192/bjp.184.5.386. PMID 15123501
- [Background] Gun SY, Titov N, Andrews G. Acceptability of Internet treatment of anxiety and depression. Australas Psychiatry. 2011 Jun;19(3):259-64. doi: 10.3109/10398562.2011.562295. PMID 21682626
- [Background] Gilbody S, Brabyn S, Lovell K, Kessler D, Devlin T, Smith L, Araya R, Barkham M, Bower P, Cooper C, Knowles S, Littlewood E, Richards DA, Tallon D, White D, Worthy G; REEACT collaborative. Telephone-supported computerised cognitive-behavioural therapy: REEACT-2 large-scale pragmatic randomised controlled trial. Br J Psychiatry. 2017 May;210(5):362-367. doi: 10.1192/bjp.bp.116.192435. Epub 2017 Mar 2. PMID 28254959
- [Background] Deady M, Choi I, Calvo RA, Glozier N, Christensen H, Harvey SB. eHealth interventions for the prevention of depression and anxiety in the general population: a systematic review and meta-analysis. BMC Psychiatry. 2017 Aug 29;17(1):310. doi: 10.1186/s12888-017-1473-1. PMID 28851342
- [Background] Christensen H, Batterham P, Mackinnon A, Griffiths KM, Kalia Hehir K, Kenardy J, Gosling J, Bennett K. Prevention of generalized anxiety disorder using a web intervention, iChill: randomized controlled trial. J Med Internet Res. 2014 Sep 2;16(9):e199. doi: 10.2196/jmir.3507. PMID 25270886
- [Background] Clarke G, Reid E, Eubanks D, O'Connor E, DeBar LL, Kelleher C, Lynch F, Nunley S. Overcoming depression on the Internet (ODIN): a randomized controlled trial of an Internet depression skills intervention program. J Med Internet Res. 2002 Dec;4(3):E14. doi: 10.2196/jmir.4.3.e14. PMID 12554545
- [Background] Cukrowicz KC, Joiner TE. Computer-based intervention for anxious and depressive symptoms in a non-clinical population. Cognit Ther Res [Internet]. Springer US; 2007 [cited 2018 Aug 3];31:677-93. Available from: http://link.springer.com/10.1007/s10608-006-9094-x
- [Background] Levin ME, Pistorello J, Seeley JR, Hayes SC. Feasibility of a prototype web-based acceptance and commitment therapy prevention program for college students. J Am Coll Health. 2014;62(1):20-30. doi: 10.1080/07448481.2013.843533. PMID 24313693
- [Background] Imamura K, Kawakami N, Furukawa TA, Matsuyama Y, Shimazu A, Umanodan R, Kawakami S, Kasai K. Effects of an Internet-based cognitive behavioral therapy (iCBT) program in Manga format on improving subthreshold depressive symptoms among healthy workers: a randomized controlled trial. PLoS One. 2014 May 20;9(5):e97167. doi: 10.1371/journal.pone.0097167. eCollection 2014. PMID 24844530
- [Background] Lintvedt OK, Griffiths KM, Sorensen K, Ostvik AR, Wang CE, Eisemann M, Waterloo K. Evaluating the effectiveness and efficacy of unguided internet-based self-help intervention for the prevention of depression: a randomized controlled trial. Clin Psychol Psychother. 2013 Jan-Feb;20(1):10-27. doi: 10.1002/cpp.770. Epub 2011 Sep 2. PMID 21887811
- [Background] Spek V, Cuijpers P, Nyklicek I, Smits N, Riper H, Keyzer J, Pop V. One-year follow-up results of a randomized controlled clinical trial on internet-based cognitive behavioural therapy for subthreshold depression in people over 50 years. Psychol Med. 2008 May;38(5):635-9. doi: 10.1017/S0033291707002590. Epub 2008 Jan 21. PMID 18205965
- [Background] Musiat P, Conrod P, Treasure J, Tylee A, Williams C, Schmidt U. Targeted prevention of common mental health disorders in university students: randomised controlled trial of a transdiagnostic trait-focused web-based intervention. PLoS One. 2014 Apr 15;9(4):e93621. doi: 10.1371/journal.pone.0093621. eCollection 2014. PMID 24736388
- [Background] Morgan AJ, Jorm AF, Mackinnon AJ. Email-based promotion of self-help for subthreshold depression: Mood Memos randomised controlled trial. Br J Psychiatry. 2012 May;200(5):412-8. doi: 10.1192/bjp.bp.111.101394. Epub 2012 Mar 22. PMID 22442102
- See also: World Health Organisation (2017) — http://www.who.int/mediacentre/factsheets/fs369/en/
- See also: Mental Health and Well being in England Adult Psychiatric Morbidity Survey 2014 — https://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment_data/file/556596/apms-2014-full-rpt.pdf